CLINICAL TRIAL: NCT05159284
Title: Prospective Evaluation of the Efficacy and Safety of Topical Hydrocortisone Treatment on Clinical Signs and Symptoms of Dry Eye Disease Associated With Moderate Meibomian Gland Dysfunction
Brief Title: Efficacy and Safety of Topical Hydrocortisone on Signs and Symptoms of Dry Eye Associated to Meibomian Gland Dysfunction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Thea, Spain (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THEA_HLF_1/21
Record Dates: First submitted 2021-10-25; First posted 2021-12-16 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: Phase IV, interventional, prospective, randomized, single blind, of parallel groups with two treatment arms clinical trial in one center.
Who Masked: Investigator
Masking Description: This is a single-blinded study for the PI or person designated to conduct the study (blinded investigator). Study medication will be labelled as blinded medication. The prescription will be done by the blinded investigator using a kit number, and study medication delivery will be done by a person designed by the PI for this topic through the study (unblinded collaborator). Patients will be instructed not to inform the investigators who perform the ophthalmological evaluation about the group they will be assigned to. Patient assessments will be performed by blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Softacort® Lephanet® Thealoz Duo® MGD Rx EyeBag®
  Interventions: Drug: Hydrocortisone Ophthalmic; Device: MGD Rx EyeBag® eyelid warming device; Device: Lephanet® lid wipes; Device: Thealoz Duo® artificial tear with trehalose 3% and sodium hyaluronate 0.15%
- Control group (Other): Lephanet® Thealoz Duo® MGD Rx EyeBag®
  Interventions: Device: MGD Rx EyeBag® eyelid warming device; Device: Lephanet® lid wipes; Device: Thealoz Duo® artificial tear with trehalose 3% and sodium hyaluronate 0.15%

INTERVENTIONS:
Drug: Hydrocortisone Ophthalmic — 1 drop 4 times daily for 12 days, followed by twice daily for 2 days and stop, for a total of 14 days of treatment. Repeat on day 28: 1 drop 4 times daily for 12 days, followed by twice daily for 2 days and stop. Patients in the intervention arm will receive two 14-day cycles of hydrocortisone.
  Other Names: Softacort®
  Arms: Intervention group
Device: MGD Rx EyeBag® eyelid warming device — Eyelid warming device used once daily for 10 minutes followed by lid massage for 12 weeks by patients in both control and intervention arm.
  Other Names: Blepha EyeBag®
Device: Lephanet® lid wipes — Lid hygiene with Lephanet® lid wipes used twice daily for 3 weeks followed by once daily for 9 more weeks by patients in both control and intervention arm.
  Other Names: Blephaclean®
Device: Thealoz Duo® artificial tear with trehalose 3% and sodium hyaluronate 0.15% — Artificial tear supplementation with Thealoz Duo® 4 times daily for 12 weeks by patients in both control and intervention arm.

SUMMARY:
The purpose of this study is assess the efficacy and safety of topical hydrocortisone (Softacort) for treatment of clinical signs and symptoms of dry eye disease when associated with moderate meibomian gland dysfunction.

DETAILED DESCRIPTION:
This is a prospective, interventional, randomized (1:1), single blind, of parallel groups and two treatment arms clinical trial (phase IV).

All patients diagnosed with dry eye disease (DED) associated with moderate MGD may participate in the study if they meet all the selection criteria.

Patients (or their representatives) will provide informed consent (IC) prior to the enrolment in the study and to the start of data collection. Patients must meet all the inclusion criteria and not meet any of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Documented diagnosis of DE defined by TBUT value ≤ 5 seconds and Schirmer I test value < 10 mm/5 min
3. Normal ophthalmic findings except dry eye disease and meibomian gland dysfunction
4. OSDI score > 23 (moderate symptoms)
5. Documented diagnosis of MGD grade 2 to 3
6. Patient who can understand the instructions and adhere to medications
7. Patient who receives complete information regarding the study objectives, authorize their participation in the study and sign an informed consent form before entering in the study

Exclusion Criteria:

1. Any contraindication or known allergies to Lephanet®, Thealoz Duo®, MGD Rx EyeBag® or Softacort®
2. Ocular surgery in the past 6 months
3. Ocular hypertension or glaucoma
4. Cicatricial MGD
5. Atopic condition including ocular allergy
6. Suspect demodex lid infestation as evidenced by the presence of collarettes
7. Intraocular inflammation
8. Confirmed infection with COVID-19 in the last 3 months
9. Systemic autoimmune disorder
10. Use of contact lenses during the month prior to inclusion in the study or during the study
11. Punctal occlusion
12. Intraocular pressure > 22 mmHg
13. Patient who has received topical or systemic anti-inflammatory treatments including corticosteroids and nonsteroidal anti-inflammatory drugs (NSAIDS) within 3 months prior to be included in the study or with a prescription for receiving topical / systemic anti-inflammatory treatments for the next 3 months
14. In the investigator´s opinion, use of systemic medications that could affect the function of the meibomian gland and tear production within 3 months prior to be included in the study
15. Any ocular or systemic disease known to affect the tear film other than MGD
16. Patient with any situation or state that in the opinion of the investigator discourages their participation in the study
17. Patient participating in any other interventional or non-interventional study or who have participated in another study within 30 days prior to inclusion in this study
18. Women who are pregnant, planning to become pregnant or breastfeeding
19. Patient who will not be able to complete the study (e.g., not willing to attend the follow-up visits, way of life interfering with compliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint: Change from baseline in Meibomian Gland Dysfunction Dry Eye symptom score (MGD-DE) at 14 days | Day 0 and Day 14
  Meibomian Gland Dysfunction Dry Eye symptom score (MGD-DE) calculated by the sum of the Visual Analogue scale (VAS) score assigned by the patient on a scale from 0 (no symptoms) to 100 (worst symptoms) in the following symptoms: itching, dry eye sensation, burning, foreign body sensation and ocular redness.
Safety endpoint: Incidence of increased intraocular pressure and change from baseline at Day 0, Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Mean of 3 measures of intraocular pressure measured with Goldmann tonometer in each eye on Day 0, Day 14, Day 28 and Day 84. Increased intraocular pressure defined as >21 mmHg.

SECONDARY OUTCOMES:
Change from baseline in Ocular Surface Disease Index (OSDI) questionnaire at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84.
  12-item questionnaire related to vision-related function, ocular symptoms, and environmental triggers of dry eye. Response on a 0 to 4 scale that ranges from "none of the time" to "all of the time". The final score is calculated by multiplying the sum of all the scores by 25 and then dividing the total by the number of questions answered. Scores range from 0 to 100 with 0 to 12 representing normal, 13 to 22 mild DED, 23 to 32 moderate DED, and 33 severe DED
Change from baseline in Meibomian Gland Dysfunction Dry Eye symptom score at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84.
  Meibomian Gland Dysfunction Dry Eye symptom score (MGD-DE) calculated by the sum of the VAS score assigned by the patient on a scale from 0 (no symptoms) to 100 (worst symptoms) in the following symptoms: itching, dry eye sensation, burning, foreign body sensation and ocular redness.
Change from baseline in ocular symptoms Visual Analogue scale (VAS) questionnaire at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  VAS score assigned by the patient on a scale from 0 (no symptoms) to 100 (worst symptoms) in each of the following symptoms: itching, dry eye sensation, burning, foreign body sensation, ocular redness, ocular fatigue, and blurry vision.
Change from baseline in hyperemia score (McMonnies-Chapman scale) at Day 14, Day 28 and Day 84. | Day 0, Day 14, Day 28 and Day 84
  Inferior conjunctival hyperemia will be estimated by comparison with the photographic conjunctival hyperemia reference scale covering six grades, with highest grade as worst hyperemia.
Change from baseline in Tear break up time (TBUT) at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film observed with slit-lamp after instillation of fluorescein. A TBUT under 10 seconds is considered abnormal
Change from baseline in corneal and conjunctival staining with fluorescein (Oxford grading scale) at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  After instillation of fluorescein in conjunctival sac a comparison to the Oxford chart panels A to E, with E being the worst outcome.
Change from baseline in corneal and conjunctival staining with lissamine green (Van Bijsterveld scale) at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Scoring system that divides the ocular surface into three zones: nasal bulbar conjunctiva, temporal bulbar conjunctiva, and cornea. Each zone is evaluated on a scale of 0 to 3, with 0 indicating no staining and 3 indicating confluent staining; the maximum possible worse outcome score with this system is 9.
Change from baseline in meniscus height at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Measured with anterior segment optical coherence tomography. The lower the tear meniscus height the worst outcome.
Change from baseline in Schirmer I test at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Folded edge Schirmer strip is placed over the rim of the lower eyelid and the eyes are then lightly closed. The amount of wetting after 5 minutes on the strip is measured in mm. Normal more than 10 mm / 5 min
Change from baseline in MGD grading at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Grading of MGD: 0 to 4 where 0 is no meibomian gland dropout and expressed meibum with clear appearance and 4 is with gland dropout of more than half the lid margin or complete keratinization of the ducts and no expression of meibum. Higher grade is a worse outcome.
Change from baseline in lid abnormalities at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Lid margin irregularity (presence or absence), thickness, and plugging of the meibomian orifices. A scale from 0 to 2, with 0 = no findings, 1 = mild findings, and 2 = severe findings.
Change from baseline in Eyelid telangiectasia score at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Eyelid telangiectasia score from 0 to 3, where 0 is no findings and 3 is severe findings.
Change from baseline in Lissamine green staining score at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Mean of longitudinal staining of upper lid margin after instilation with lissamine green graded from 0 to 3 and sagittal staining graded from 0 to 3 estimated by comparison with standard chart. Higher grade is a worse outcome.
Change from baseline in Meibomian gland expressibility score at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Express each of 5 glands in temporal, central and lower lid and grade each gland on a scale from 0 to 3, with 3 = clear liquid secretion, 2 = cloudy liquid secretion, 1 = inspissated / toothpaste consistency, and 0 = no secretion. Total score range from 0 to 45. A lower grade is a worse outcome.
Change from baseline in tear inflammatory cytokines at Day 14 | Day 0 and Day 14.
  Levels of 8 inflammatory cytokines in tears will be determined 2 micro liter samples taken from each eye.
Incidence of adverse events and serious adverse events occurred during the study. | Day 0, Day 14, Day 28 and Day 84
  Report of any untoward medical occurrence in a patient during the study
Change from baseline in ETDRS visual acuity at Day 14, Day 28 and Day 84 | Day 0, Day 14, Day 28 and Day 84
  Best corrected visual acuity in each eye measured with the ETDRS optotype.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Hervas Ontiveros, Dr, Principal Investigator — anheront@gmail.com
Locations (1):
- Hospital La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No